CLINICAL TRIAL: NCT02275715
Title: Treatment of Feeding Problems in Children With Autism
Acronym: PT-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Rochester (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400831-N
Record Dates: First submitted 2014-10-15; First posted 2014-10-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Treatment of Feeding Problems in Children With ASD
Keywords: autism spectrum disorder (ASD); feeding problems
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Training Program (PT-F) (Experimental): Treatment group
  Interventions: Behavioral: Parent Training Program
- Waitlist (No Intervention): Control group in which parents randomized to this group will be offered the PT-F at the end of the 20 week study period to address their child's feeding issues.

INTERVENTIONS:
Behavioral: Parent Training Program — An 11-session manualized behavioral parent training program for the treatment of feeding problems teaching parents to use a range of behavioral procedures to address a variety of common feeding problems.
  Other Names: PT-F
  Arms: Parent Training Program (PT-F)

SUMMARY:
The primary aim of the project is to develop and pilot a manualized, individually delivered Parent Training Program for Feeding Problems (PT-F) in children with autism spectrum disorder (ASD) to assess feasibility and parent acceptance of the program. The secondary aim of the project is to assess the success of the PT-F program in improving mealtime behavior problems when compared to the wait-list control.

Exploratory aims include obtaining preliminary data on the impact of PT-F on child and parent functioning (reducing parent stress and improving parent sense of competency and parent-child interactions at mealtime), assessing the impact of treatment on interfering behaviors around mealtime/snack times, and measuring nutritional improvements after treatment.

DETAILED DESCRIPTION:
Fifty well characterized children will be randomly assigned to either the 20 week PT-F or a waitlist control group. Study assessments evaluating feeding and mealtime behaviors, nutritional intake, daytime behaviors, repetitive behaviors, sensory sensitivities, parent stress and parent-child interactions will be completed at Baseline, Week 10, and Week 20 timepoints. Treatment Fidelity forms will be completed by the therapist at the end of each treatment session to assess achievement of session goals and parent adherence during each session.

ELIGIBILITY:
Inclusion Criteria

1. Males and females >=2 and < 8 years of age.
2. At least one participating parent resides with the child >50% of time.
3. Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnosis of Autism Spectrum Disorder as established by clinical assessment, corroborated by the Autism Diagnostic Interview - Revised (ADI-R) and Autism Diagnostic Observation Schedule - 2nd Edition (ADOS2).
4. A total score of > 54 on the Brief Autism Mealtime Behavior Inventory. A score of 54 is one standard deviation above the mean for the ASD group, as reported by the developers.
5. A receptive language level of 12 months or greater. [Rationale: diagnostic uncertainty of ASD in children functioning below 12 months of age and the need for the child to understand simple instructions in PT-F].
6. Medication free or stable medications and/or supplements (no changes in past 6 weeks and no planned changes during study period). [Rationale: Many children with ASD are on medications to target associated behaviors. These include stimulants and atypical antipsychotics. Excluding these children could result in a non-representative sample of children with ASD and feeding problems. We will require that the feeding problems pre-date the initiation of medications / supplements].

Exclusion Criteria

1. Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnosis of Rett's Disorder or Childhood Disintegrative Disorder.
2. Presence of a known serious medical condition in the child influencing the management of diet and treatment impacting diet or appetite (e.g., current or past gastroesophageal reflux disease, significant food allergies, diabetes, cystic fibrosis, celiac disease, endocrine disorder, genetic disorders known to impact growth or appetite). [Rationale: these children may require different treatments than the behaviorally based parent training intervention].
3. Significant oral motor dysfunction (i.e., unable to safely chew and swallow age appropriate textures).
4. Presence of known psychiatric diagnosis in the child that would require a different treatment (e.g., psychotic disorder, major depression).
5. Inpatient hospitalization.
6. Being fed via nasogastric or gastrostomy tube in the past year.
7. On medication or supplements specifically targeting appetite.
8. Insufficient proficiency of English language prohibiting comprehension of PT-F. [Rationale: Parents will need sufficient command of English to benefit from the English materials].

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Complete Data | Week 20
  Measure of feasibility of randomized controlled trial by successful recruitment of 50 subjects with complete data collected from > 80% (> 40) subjects.
Treatment Fidelity | Week 20
  Measure of therapists' ability to deliver PT-F with > 80% average fidelity as rated by fidelity checklists
Parent Adherence | Week 20
  Measure of parent adherence to the intervention as evidenced by average attendance of > 80% of scheduled sessions and successful completion of > 70% of session activities as rated from adherence checklists.

SECONDARY OUTCOMES:
Brief Autism Mealtime Behavior Inventory (BAMBI) | Baseline, Week 10, Week 20
  Measure of mealtime behavior problems

OTHER OUTCOMES:
Parent Functioning | Baseline, Week 10, Week 20
  Measure of parent reported stress, competency, and parent-child interactions at mealtime as rated by the Parenting Stress Index, Caregiver Strain Questionnaire, Parenting Sense Of Competence, and About Your Child's Eating
Interfering Behaviors at Mealtime | Baseline, Week 10, Week 20
  Measure of repetitive behaviors, sensory sensitivities, tantrum, irritability, and noncompliance as rated by the Repetitive Behaviors Scales - Revised, Short Sensory Profile, Aberrant Behavior Checklist, and Home Situations Questionnaire
Healthy Eating Index | Baseline, Week 10, Week 20
  Measure of nutritional intake

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Johnson, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Rochester, Rochester, New York